CLINICAL TRIAL: NCT03019341
Title: Immediate Nausea and Vomiting After the Administration of Non-ionic Contrast Media: Prevalence and Risk Factors
Brief Title: Immediate Nausea and Vomiting After the Administration of Non-ionic Contrast Media
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Soon Ho Yoon, Assistant professor, Department of Radiology, Seoul National University Hospital, Seoul National University Hospital
Other Study IDs: SeoulNUH_NVICM
Record Dates: First submitted 2016-12-31; First posted 2017-01-12 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Contrast Agent; Nausea
Keywords: Nausea; Vomiting; Non-ionic contrast media; Side effect
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with enhanced CT scan: Patients undergo CT examination after the administration of non-ionic contrast media for clinical need.

SUMMARY:
The prevalence of nausea and vomiting after the administration of non-ionic contrast media has rarely been assessed. Thus, the aim of our study is to evaluate the prevalence and risk factors of nausea and vomiting after the exposure to the non-ionic contrast media for computed tomography examinations in adults.

DETAILED DESCRIPTION:
There is no robust evidence or guideline for fasting prior to contrast-enhanced CT scan in patients. Substantial heterogeneity exists on fasting prior to contrast-enhanced CT worldwide. Through dedicated questionnaires, the investigators plan to prospectively assess the prevalence and the risk factors for nausea and vomiting after the exposure to the non-ionic contrast media agent in adult patients undergoing computed tomography examinations.

ELIGIBILITY:
Inclusion criteria:

* Patients undergoing contrast-enhanced CT examination with non-ionic contrast media during regular working hours
* Adult patients (20 years old or older)
* Patients with informed written consent
* Patients under observation by medical staffs during and after CT examination up to 30 minutes.

Exclusion criteria:

* Patients without informed written consent
* Age of patients younger than 20 years old
* Uncooperative patients
* Pediatric, pregnant, and emergent patients
* Patients without sufficient observation by medical staffs during and after CT examination up to 30 minutes.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo elective CT examination after the administration of non-ionic contrast media in a single tertiary hospital will be enrolled based on following inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 1175 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of immediate nausea or vomiting after contrast injection | For 30 minutes after administration of non-ionic contrast media
  Patients will be observed for 30 minutes after the administration of the contrast media agent and medical staffs will record and evaluate the patients' status and the severity of gastrointestinal reaction to the contrast media agent such as nausea or vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Soon ho Yoon, Study Chair — Seoul National University of Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee BY, Ok JJ, Abdelaziz Elsayed AA, Kim Y, Han DH. Preparative fasting for contrast-enhanced CT: reconsideration. Radiology. 2012 May;263(2):444-50. doi: 10.1148/radiol.12111605. PMID 22517959
- [Background] Federle MP, Willis LL, Swanson DP. Ionic versus nonionic contrast media: a prospective study of the effect of rapid bolus injection on nausea and anaphylactoid reactions. J Comput Assist Tomogr. 1998 May-Jun;22(3):341-5. doi: 10.1097/00004728-199805000-00001. PMID 9606371